## Peanut/Tree Nut Desensitization and induction of tolerance in Children

#### 1 Proposed Research Questions

- 1. What is the rate of desensitization in children allergic to peanuts or tree nuts?
- 2. Is the efficacy of a maintenance protocol of 300mg peanut protein similar to the efficacy of a maintenance protocol of 30mg peanut protein?
  - 3. What are the predictors associated with success or failure of desensitization in children?
  - 4. What are the molecular mechanisms involved in desensitization to peanut/tree nut?

## 2 Research Objectives and Significance

The investigators are proposing to initiate a study assessing a common desensitization protocol for peanut/tree nut allergy

This study would enable us to better determine the potential benefit of desensitization in individuals with peanut/tree nut allergy.

More specifically, the investigators will address the following research objectives:

#### **Objectives**

- A. To develop a protocols for peanut/tree nut desensitization with high (300mg) and low (30mg maintenance dose).
  - B. To determine the rate of desensitization to peanut/tree nut.
  - C. To characterize predictors of successful desensitization.
  - D. To characterize molecular mechanisms involved in the process of desensitization.

#### 3. Gaps and Unmet Needs in Existing Knowledge on food desensitization

# 3.i Why do the investigators need trials on food desensitization.

Foods are reported to be primary inciting allergens for anaphylaxis and account for 33.2% to 56% of all anaphylaxis cases. (1-4) Further, food-induced anaphylaxis hospital admissions are reported to have increased, mainly in the first 2 decades of life. (5;6)

At present, the only treatment for food allergy is to avoid the allergy-causing food, while the only treatment for an allergic reaction is prompt administration of intramuscular epinephrine. (7;8)

Primary anaphylaxis prevention is based on allergen desensitization through immunotherapy and until recently was not available for food allergies. Although there are a few recent research protocols exploring desensitization for foods and although these have so far been largely successful, <sup>(9;10)</sup> up to this point there are no known guidelines describing the optimal candidate for desensitization nor are there criteria for the safest and most effective dosing schedule. Further, many of these studies have a very small sample size and do not use a control group. Hence, the efficacy of these protocols is hard to interpret <sup>(11-14)</sup> and additional larger scale randomized control studies are required.

# 3.ii Why peanut/tree nut.

Peanut and tree nut allergies are the most common food allergies in children and adults in Canada affecting almost 2% and 1.5% of the population respectively. (15) and recent reports suggest that only 10%-20% will out-grow nut allergy. (16)

Further, peanut and tree nut allergy are most common trigger for anaphylaxis and the most common trigger for recurrent anaphylaxis. (17)

With the support of AllerGen NCE and CIHR the investigators have initiated in 2014 the first cross Canada study to assess desensitization to milk. This study now includes

almost 50 patients, and our preliminarily results reveal an almost 80% success rate. In April 2016 in collaboration with Aimmune the investigators have initiated the first oral desensitization to peanut. (18) The investigators are now proposing to develop a protocol for peanut and tree nut desensitization based on the expertise, recruitment skills and data collected in our first 2 years of milk desensitization and more recently peanut desensitization.

Peanut and tree nuts are the most common foods causing acute allergic reactions and almost all fatal reactions in North America had been triggered by peanutor tree nuts. The term "tree nut" is collectively used to categorize nuts that grow on trees. Prevalence of individual tree nut allergies varies significantly by region, with hazelnut being the most common tree nut allergy in Europe, walnut and cashew the most common in the USA and Brazil nut, almond and walnut most commonly reported in Europe. (19) In Canada alone, recent research has shown up to 2% of children and 1% of adults have peanut allergy. (15;21)

The main peanut allergens are Arah1 and Arah2 .<sup>(22)</sup>Mosttree nut allergens identified to date are seed storage proteins such as the vicilins, legumins, americ globulins, and 2S albumins. Othertree nut allergens include profilins and hevein- related proteins, known for their contribution to the allergenicity of a wide variety of pollens, nuts, seeds, fruits and vegetables and their propensity for exhibiting a significant degree of IgE- mediated cross- reactivity. <sup>(23)</sup> Cross-reactivity among nuts may occur because of minor constituent panallergens such as profilins and lipid transfer proteins, or may involve major nut storage protein allergens, including albumins, legumins, and vicilins. <sup>(24)</sup>Strong cross-reactivity was present among walnuts, pecans, and hazelnuts, and mild cross- reactivity was present among cashews, Brazil nuts, pistachios, and almonds. <sup>(202)</sup>
Diagnosis of peanut/tree nut allergy is confirmed by having a convincing clinical history as well as the presence of a positive SPT defined as a wheal diameter at least 3 mm larger than that elicited by the negative control within 10 to 15 minutes of placement, provided

by a physician, or an IgE level of at least 0.35 KU/L. (25) If however, exposure to

peanut/tree nut never occurred, or if clinical history is uncertain, diagnosis is based on having a positive SPT and a tree nut- specific IgE above 15 kU/L. (26)

Despite the importance of peanut and tree nut allergy, there are only three studies assessing oral immunotherapy for peanut and there is only one group that published to date a research desensitization to hazelnuts. No protocols have been published so far for other tree nuts. The protocol for hazelnuts reveals encouraging results with significantly increased thresholds to food induced allergic reactions after oral immunotherapy in the majority of those with hazelnut allergy<sup>(18;27;28)</sup> In conclusion, the efficacy of the immunotherapy, extent of desensitization versus tolerance, the quantity/ frequency of allergen consumption required to maintain this effect and molecular mechanisms involved in the desensitization process are currently unknown.

# 3. iii. Do the investigators achieve only desensitization or do the investigators induce also tolerance.

Desensitization refers to a change in the amount of food antigen needed to cause allergic symptoms; this state is dependent on regular antigen exposure. In contrast, *tolerance* refers to long-term immunologic changes associated with the ability to ingest a food without symptoms and without ongoing therapy. Desensitization is a worthwhile therapeutic goal as it allows individuals freedom from the risk of accidental ingestion in everyday settings; achieving long-term clinical tolerance would allow safe food ingestion without ongoing therapy by inducing lasting immunologic changes. Trials so far suggest that might be loss of tolerance within 48 h after elimination of the food from the diet. However, these trials are flawed by their small sample size (3 patients). In a recent study it was reported that prolonged (at least 4 years) daily immunotherapy is

crucial for achieving Sustained Unresponsiveness (SU)=lack of dose limiting symptoms during DBPCFC and also 4-6 weeks after stopping OIT. (31)

#### 3. iv Gaps related to the appropriate maintenance dose of peanut desensitization.

The threshold doses of peanut and tree nut that trigger reactions ranges from 15 mg to 1000mg <sup>(32-34)</sup> and studies suggest that almost a third of products from Western Europe and two thirds of products from eastern Europe without precautionary labeling contain detectable levels of peanut or tree nut protein up to 245 mg per liter. <sup>(35)</sup> Hence it is crucial that desensitization protocols will be efficacious in protection against reactions to at least 300mg of peanut or tree nut protein. One previous study on peanut had shown similar efficacy in attaining sustained unresponsiveness (defined as no allergic reaction to 5 g of peanut ingested 1 month after stopping oral immunotherapy) between a protocol with 3000 mg maintenance dose versus 300mg. <sup>(36)</sup> .It is of crucial importance to assess the efficacy of low dose protocols as trials aiming for high doses of peanut maintenance are associated with up to 40% drop-out due to adverse effects .

#### 3.v Gaps regarding the roles of mast cells in desensitization.

Given that food desensitization is a relatively rapid process, mast cell are implicated to have a key role in this process. Compared to activated cells, desensitized Mast cells were shown to have had impaired degranulation, calcium flux, secretion of arachidonic acid

products.<sup>(37)</sup> However, the effect of food desensitization on mast cells was not explored so far in clinical trials.

## 3vi. Gaps regarding the role of T regulatory cells in desensitization.

Although several studies in humans report that food allergens induce specific effector T cells, there are significant controversies between studies regarding the T cell phenotype dominating that response. Some studies report a Th2 dominated response in children with food allergies whereas Th1- responses underlie oral tolerance (38). Other studies suggest that food antigens induce a Th2 response regardless of the presence of food allergy (39). Further, it is proposed that Treg cells may be crucial to control food related allergic reactions. A potential suppressive role of Treg in food allergies was exemplified in both animal models (40-42) and in human studies. Increased numbers of Treg cells in peripheral blood in children who outgrew allergy was reported (43,44) and decreased Treg suppression was associated with allergy in neonates (45). Cord blood from offspring of atopic mothers showed fewer innate induced Treg cells and impaired supression (46). In line with these, an association with severe food allergy was described in patients with profound dysfunction of T reg cells that characterizes IPEX syndrome (immunodysregulation polyendocrinopathy enteropathy X-linked syndrome)

In contrast 1 study looking at the number of Tregs in 10 children undergoing desensitization reports no enhancement of CD4+CD25+Foxp3+ T(reg) levels in peripheral blood and suggests that there is unlikely a role for long-lasting systemic immunologic changes in desensitization. However, this study is limited by a small sample size and relatively short period of follow up (6 months). (48)

#### 3.vii Gaps regarding the role of demethylation in desensitization.

The rising incidence of food allergies is occurring more rapidly than changes to the genome sequence would allow<sup>(49)</sup> and recent studies suggest that epigenetic regulation (heritable changes in gene expression that occur in the absence of alterations in DNA sequences) may in part mediate the complex gene-by-environment interactions that can lead to asthma.<sup>(50)</sup> Experimental studies provide substantial in vitro data indicating that

DNA methylation of genes critical to T-helper cell differentiation may induce polarization toward or away from an allergic phenotype. Methylation of DNA and resulting changes in chromatin structure have been shown to initiate the process by which the Th cells lose their plasticity and differentiate productively toward the Th1 versus the proallergic Th2 pattern of cytokine gene expression. (51-53) So far no studies have explored the role of DNA methylation in short term processes such as desensitization for food allergens.

## 3viii Effect of Heat Treating Peanuts/Tree Nuts on Allergenicity

There is ample evidence in the literature that there is a significant increase in the allergenicity of peanuts after undergoing thermal processing (i.e. roasting). Glycation at high temperatures via the Maillard reaction, the addition of amines on reducing sugars to provide Schiff bases and advanced glycation end products (AGEs), is proposed to be the primary mechanism of enhancement of allergic responses in roasted peanuts. Our primary objective is to develop strategies to decrease glycation and Maillard reaction products in the thermal processing of peanuts.

We propose to use High-Resolution Magic Angle Spinning Nuclear Magnetic

Resonance Spectroscopy (HR-MAS NMR) to take an array of molecular snapshots of

intact raw peanuts from room temperature to roasted temperatures (i.e. 20-150°C) and to subsequently perform an antigen-specific ELISA, which measures IgE binding, to assess the allergenicity at each temperature. We will expand the approach to variable temperature studies under conditions where small molecules, such as sugars and amino acids, are removed from intact or macerated peanuts prior to heating.

## 4. Methodological Approach/Study Design

Seventy five males and females between 2 to 40 years of age, diagnosed with peanut /tree nut allergy will be approached by our study group. Participants will be recruited from the allergy clinic at the Montreal Children's Hospital and at collaborating sites in Toronto and Vancouver Participants who meet inclusion criteria will be enrolled in a desensitization programme specific to their allergy. Thus a peanut allergic participant will be desensitized to peanut only, while a patient allergic to cashew for example, will be desensitized to cashew only. Patients with more than one peanut or nut allergy will be offered the choice of to which allergen they would prefer to be desensitized

**Inclusion criteria:** Children and adults between 2 and 40 who satisfy all the following criteria will be included:

• A history suggestive of immediate allergy to peanut/tree nut. A convincing clinical history of an IgE mediated reaction to a specific food will be defined as a minimum of 2 mild signs/symptoms or 1 moderate or 1 severe sign/symptom that was likely IgE mediated and occurred within 120 minutes after ingestion or contact (or inhalation in the case of fish and shellfish).

Reactions will be considered mild if they involve pruritus, urticaria, flushing,

or rhinoconjunctivitis; moderate if they involve angioedema, throat tightness, gastrointestinal complaints, or breathing difficulties (other than wheeze); and severe if they involve wheeze, cyanosis, or circulatory collapse. (54-57)

- The presence of at least one of the following confirmatory tests:
  - Positive SPT to peanut/tree nut or its proteins (weal diameter 3 mm larger than that of the normal saline control). The allergens used will be commercial extracts of peanut/tree nut (Omega Labs, Toronto, Ontario).
  - Detection of serum specific IgE (>0.35 kU/L) to peanut/tree nut or any of its proteins, measured by fluorescence enzyme immunoassay (Phadia, CAP System, Uppsala, Sweden).
  - Positive oral challenge test to peanut/tree nut. Oral challenges will be performed with raw peanut/tree nut according to the recommendations of the position paper of the European Academy of Allergology and Clinical Immunology (58).
- Informed consent form signed by the parents or legal guardian (appendix B).

## **Exclusion criteria.**

- Patients who are unstable from a respiratory point of view ...
- Patients who present with intercurrent disease at the time of starting desensitization.
- Non-IgE-mediated or non-immunological adverse reactions to nuts.

- Malignant or immunopathological diseases and/or severe primary or secondary immune deficiencies.
- Patients receiving immunosuppressor therapy
- Patients receiving β-blockers (including topical formulations).
- Associated diseases contraindicating the use of epinephrine: cardiovascular disease or severe hypertension.
- Patients diagnosed with eosinophilic gastrointestinal disorder.

#### **STUDY PROCEDURES**

The desensitization protocol will be performed at the Center of Innovative medicine (CIM) as is currently done for our peanut desensitization study, under the direct supervision of the medical and nursing staff, and with full cardiopulmonary resuscitation measures available for the treatment of possible allergic reactions that could occur during the procedure. Oral and intravenous doses of diphenhydramine and intramuscular epinephrine were at the bedside at all times.

# Desensitization to peanut (B1 and B2).

# **Oral Food Challenge**

Patients will begin with a blinded, placebo-controlled oral food challenge (BPCFC) to peanut that will take place over two days, with patients receiving doses of placebo one

day and peanut/tree nut protein the other. In all cases, protein will be in the form of crushed peanut/tree nut. All challenges and desensitization procedures will be done with commercially available peanut/tree nut proteins. Patients and evaluating physicians will be blinded, but not the study nurses nor the study coordinator. On both days, patients will arrive at the Center for Innovative Medicine (CIM) in the morning. The CIM services include equipment and medications required to monitor and treat potential reactions. The CIM nurse that will assist in the desensitization protocol is a nurse that has been trained to work in an intensive care unit. Patients will be reminded beforehand that they must be in good health for the challenge. If they are not in good health, the challenge will be rescheduled. Upon arriving, a physical exam will be performed and vital signs taken. Skin prick test to peanut/tree nut will be performed to establish baseline values in both. An IV catheter will be inserted in the patient's arm. The doses will be mixed in a food vehicle tolerated by the participant, such as pudding or fruit puree, that the participant is known to tolerate. Doses will be given by the study nurse every 15-20 minutes, depending on patients' tolerance of the dose (see Appendix B for challenge doses). If participants tolerate the last, 300 mg dose, they will be given a dose of food that contains the allergen in question – peanut butter in the case of a peanut challenge. Nutella in the case of hazelnut allergy. The study nurse will be with the participant for the duration of the challenge and as soon as the participant demonstrates objective signs of an allergic reaction, the challenge will be stopped and the reaction treated. Participants will be kept under observation in the CIM for two hours after the resolution of the last symptoms.

Given the similarity of allergens between walnut and pecan and cashew and pistachio (202), the investigators will offer challenge with the two cross reacting allergens (1 week to 4 weeks apart) for participants who report an allergy to at least one of these allergens.

#### Randomization

Through a process of stratified randomization (according to sex), participants will be randomly assigned in a 1:1:1 fashion to one of 3 study groups. The first group: group A will receive active desensitization with a maintenance dose of 300 mg, the second, group B will receive active desensitization with a maintenance dose of 30 mg, and the third group C group will not receive any treatment but will be followed up regularly (appendix B protocols). Patients in groups A and B will be blinded to their group assignment. Participants randomized to group C will be offered the opportunity to enter the desensitization programme after their year of observation ends. They will be randomized in a 1:1 fashion to either the 300 mg protocol or the 30 mg protocol.

## **Rush Desensitization**

The investigators will base our proposed desensitization protocol on previous studies by our group on a peanut desensitization protocol that has been active in the last year at the Montreal Children's Hospital. The modified rush two days will begin with a first single dose of 0.5 mg of peanut/tree nut protein. After the initial dose, subjects will receive approximately doubling doses every 30 minutes until a dose of 5 mg. All doses will be mixed with an acceptable vehicle food chosen by the subject and his or her parent. Those who tolerate 5 mg, will be asked to return the next day for one dose of 3 mg. If

this is tolerated, participants will be supplied with enough peanut/tree nut protein to be able to take a daily dose of 3 mg for the following 2 weeks and will come to the Montreal Children's hospital after at the end of these two weeks for a dose of 6 mg (doses will be aliquoted and put in capsules by a professional pharmacist).. Self-administered epinephrine will be provided to all patients' caregivers, along with instructions and indications for administration and education about the nature of possible reactions to OIT. Patients who are unable to complete the rush desensitization will not be eligible to continue the study

Successful desensitization will be defined when the patient will be able to tolerate 300mg of peanut/tree nut protein. A slow regimen will be used in those patients who will experience repeated moderate reactions or any severe reaction to a given dose; that regimen will consist of reducing the dose to the previously tolerated dose for 1-2 weeks or splitting the dose into two equal portions according to the discretion of the PI or co-PI.<sup>(11)</sup>

SPT with the allergens listed above will be performed on all patients before starting desensitization, and the tests will be repeated at 3, 6 and 12 months. Blood tests will be also performed to measure sIgE and sIgG, T cell phenotypes (including regulatory Tcells), vitamin D levels and DNA methylation before desensitization, at 3 weeks and at 3, 6 and 12 months.

Reactions during the desensitization protocol will be classified according to the categories proposed by Perry et al.<sup>(59)</sup>: mild reactions are defined when symptoms are limited to the oral mucosa or the skin; severe reactions include cardiovascular or

respiratory symptoms or involvement of any four systems; all other reactions will classified as moderate, although the investigators will consider isolated abdominal discomfort as mild when it lasted for 30 min or less.

The protocol will be individualized according to each patient's tolerance to peanut/tree nut:

- Mild allergic reactions will be treated when necessary and the regimen will be continued when the patient becomes asymptomatic. The previously tolerated dose will be repeated before resuming the process.
- Moderate reactions will be treated and desensitization would be restarted on the following day at the previously tolerated dose.
- Severe reactions will be treated with the necessary measures and in the appropriate department, followed by an assessment of whether to interrupt desensitization or reduce the dose on the following day to 1/10 of the dose that caused the reaction.

## **Build-up phase**

Two weeks after the two-day rush Desensitization, participants will begin the build-up phase. Participants will come to the CIM every two weeks to receive their first dose at each level. Participants will then consume this dose at home for two weeks, then return to the CIM for the next dose augmentation (doses are listed in Appendix B). Home doses will be provided in individual preweighed containers, and subjects will be instructed to ingest 1 dose daily for 2 weeks. Dose escalations will be made at visits in the research unit to ensure that subjects tolerate increases, and subjects will be observed for at least 2 hours after increases for signs of clinical reactions. This process will be repeated for 11

doses (22 weeks) with almost doubling of the dose in each hospital visit till a dose of 300mg is reached for group A. For group B participants will attain 30 mg after 6 weeks and will continue with the same dose for 16 weeks

#### Follow-up / Maintenance phase

In order to compare the efficacy of a 30 mg peanut protein dose to that of a 300 mg dose in inducing peaquat/tree nut desensitization, participants in Groups A nd B will both undergo DBPCFC at similar time points during the maintenance phase. The first of these challenges will take place one year after beginning desensitization. Participants in either group whose progress is delayed because of symptoms during the escalation phase will undergo their DBPCFC three months after attaining their maximal dose (either 30mg or 300mg). The subjects will be also instructed to otherwise continue a peanut/ tree nut-elimination diet for the duration of the study.

Subjects and families will be asked to complete daily home diaries to document that daily doses were taken, as well as to report accidental ingestions, problems with dose administration, or related symptoms. Follow-up visits in addition to or in conjunction with the biweekly visits for dose escalation will be planned at 3, 6, 9, 12 months from enrollment. Each visit will involve a medical history and physical examination. SPT, serum tree nut-specific IgE and IgG concentrations, T cell penotyping and DNA methylation will be measured at enrollment and at follow-up visits. At the 9-month follow-up visit, subjects from both groups will undergo another DBPCFC, similar to that done following escalation.

The patients' parents will be instructed verbally and in writing about the recommendations to be followed after desensitization and how to treat possible allergic

reactions. They will also given a direct telephone line to members of the study staff for consultation. Patients will be told not to perform physical exercise <sup>(60;61)</sup> for 2 h after eating and not to take non-steroidal anti-inflammatory drugs for 3 h before or after ingestion. No special recommendations will be given for viral infections.<sup>(11)</sup>

#### Food challenges

As indicated above, subjects who tolerate 300mg (group A) or 30mg (group B) of peanut/tree nut will have a two more BPCFC to determine their allergenic reactivity to peanut protein. The first of these challenges will take place one year after they begin desensitization. Participants in either group whose progress is delayed because of symptoms during the escalation phase will undergo their DBPCFC three months after attaining their maximal dose (either 30mg or 300mg). . Subjects will continue OIT dosing through the day before the challenge. One challenge will consist of doses of peanut/tree nut protein given every 10 to 20 minutes starting at 1 mg in increasing amounts up to a total of 2044mg of peanut/tree nut protein (See Appendix B, section A1 for doses). The other challenge will consist of placebo given also in 6 doses. All negative challenge results will be confirmed by means of open challenge, with at least three peanuts/tree nuts provided 1 hour after completion of the double-blind portion. The second DBPCFC will take place nine months into the Follow-Up/ Maintenance phase. Participants who pass these challenges will be instructed to continue to ingest the maintenance dose daily to the end of the follow-up period.

Participants in Group B who have allergic reactions during this oral food challenge will re-entered into the Escalation Phase and proceed to the 300 mg dose.

At the end of the study, oral desensitization will be offered to the control patients who had not achieved tolerance.

Participants who had challenges to both cashew and pistachio will repeat the challenges to both nuts at this time point. This will be done to assess whether desensitization to one of these nuts confers protection to the other, antigenically-similar nut

**Variables measured.** The following variables will be measured in each patient:

A. The primary study variable will be the presence of desensitization defined by the ability to toleratepeanut/tree nut 1 year after the start of the trial. This is a qualitative variable with three categories: total desensitization ( 300mg of peanut/ nut protein); partial desensitization ( 30-300mg of peanut/ nut protein); and failed desensitization (<30 mg of peanut/ nut protein). Only patients presenting total desensitization will be regarded as being successfully desensitized.

- B. Secondary variables will be:
- 1. Number and severity of adverse reactions occurring after oral exposure topeanut/tree nut during the desensitization and follow-up phases.
- 2. Minimum dose of peanut/tree nut that triggered symptoms during the desensitization protocols or challenge tests.
  - 3. Days until desensitization was achieved, excluding weekends.
  - 4. Indices of desensitization:

SPT weal size and levels of sIgE and sIgG before desensitization, during follow-up and at the end of the study.

#### 5. Mast cell activation.

Mast cell activation will be assessed through a proxy measure: the basophil activation test. This test is based on the percentage of CD63-expressing basophils detected by flowcytometry. This test is done by incubating basophils from highly sensitized atopic donors or preferably after priming them with Il-3 (regardless of basophil source) (62;63) with sera from patients. The investigators will assess the expression of CD63 on basophiles after addition of tree nut/antigens respectively as well as an irrelevant antigen (gliadin and tetnus toxoid) The expression of CD63 on these cells is compared to values acquired after incubation with healthy controls and the same antigens. Values above the mean of CD63+ cells + 2 SD induced will be considered as positive. (64)

#### 6. Indices of T cell tolerance:

Levels of Treg and cytokine release at base line and during desensitization. In order to characterise molecular pathways associated with desensitization, the investigators will draw 5 cc of blood from each participant and check their T cell phenotype including their Treg cells and the response to peanut/tree nut protein. As control the response to an irrelavent antigen (gliadin) and to tetanus toxoid will be assessed. The investigators will invite participants for annual follow ups in the first 5 years after study entry. The investigators will also offer the desensitization to the control group at the end of the study.

7. Health-Related Quality of Life (HRQL) can be measured in food allergy and was validated for both children and adults. (65;66) Given that HRQL measurements may be used to measure the effects of an intervention on the patient's quality of life,

patients will be asked to fill a validated HRQL for children (up to 18 years) $^{(65)}$  at study entry and after completing 12 months of maintenance

#### 5. Statistical Considerations

Given that previous studies in adults have attributed at least 50% improvement in the ability to tolerate peanut/tree nut,  $^{(67)}$  with an  $\alpha$  of 0.05 and a power (1-  $\beta$ ) of 0.80, a sample of 17 cases for group A , 17 for group B and 17 controls will be recruited. Statistical analyses will be performed using paired t-tests. A P value of <0.05 will be considered significant.

Descriptive statistics of the variables including means, standard deviations and frequencies will be computed for all study variables. The concentrations of-sIgE and sIgG, the weal size, Mast cell, T cell and DNA methylation status **and HQRL scores** at the different study time-points will be compared with their baseline values using the one-sample paired t-test, and to the control using a 2 sample t-test.

Multiple regression models will be used to assess factors associated with response to desensitization (i.e. baseline demographic characteristics; gender; age; baseline basophile activation; T cell status, baseline SPT and specific IgE, DNA methylation status, vitamin D status and season).

#### 6. Ethical Considerations

In the consent form given at study enrolment, participants will be advised that they will be randomly assigned to either desensitization treatment or observation alone for one year, (appendix B). Participants will also be advised that their data will be shared only among the study members. Participants who will be at the control group will be told that they will be offered the desensitization protocol one year after study entry.

## 7. Confidentiality and Data Management

All research documents (case report forms, questionnaires, etc) will be stored in a locked cabinet in the Centre for Innovative Medicine (CIM) at the Glen. This facility has limited access, such that non-research personnel cannot access the area.

Electronic study records will be kept on a password-protected computer in the CIM.

All participants will be assigned a unique study number and study information will be entered under this study number. The key linking the participant and their study number will be kept by the principal investigator.

Once the study has been completed, all physical study documents will be archived for 25 years at Iron Mountain. Electronic information will be stored by the Principal Investigator for 25 years

#### 8. Research Deliverables and Milestones

| Timeframe | Deliverables | Milestones |
|---|---|---|
| 08/16 – 03/ 17 | Develop sampling frame; ethics approval; | Ready to recruit participants |
| 05/17 -08/19 | Collect data from participants | 12 weeks of data collection in |

treated participants completed

08/19– 12/23 Knowledge translation activities:

Preparation of abstracts and

dissemination workshops & manuscript

manuscript

preparation

# 9. Requirement for networking across Disciplines and Sites

Our researchers have a legacy of working across disciplines, across sites, and across sectors. For this study, the investigators have assembled a multi-institutional research team with cross-disciplinary expertise Dr Ben-Shoshan (Montreal Children's Hospital, McGill University) and Dr Mazer and Dr McCusker (Montreal Children's Hospital) bring expertise in clinical immunology to the research team. Dr. Ann Clarke (Montreal General Hospital) will bring expertise in the field of clinical allergy and together with Dr. Ben-shoshan, will assisted with the study design and will supervise the statistical analyses. Epidemiologic and biostatistician skills are essential to undertaking this program of research and are represented in the persons of Moshe Ben-Shoshan (McGill) Msc in Epidemiology and Mr. Duncan Lejtenyi. Mr Duncan Lejtenyi will also be responsible for the laboratory evaluation of CD63 levels. Finally, as incorporated in our protocol, the investigators will share the results of this research with representatives of key constituencies involved in the data collection –patients with food allergies and

their families, physicians and allied professionals (e.g. nurses) through scientific meetings, our the investigators being and publications in medical journals.

# 10. Organization of Research Team

The nominated principal applicant, Dr. Moshe Ben-Shoshan, and co-principal applicants, Dr. Bruce Mazer, will oversee all aspects of the proposed research. The collaborators, Dr Stark, Dr Piccirillo and Dr Bar-Or will aid in the recruitment of patients and the assessment T cells and DNA methylation status respectively. Dr Julia Upton from Sick Kid's Hospital in Toronto and Dr Edmond Chan at BC Children's Hospital are external collaborators and will recruit patients from their respective centers Mr Duncan Lejtenyi, who had worked with our team in numerous studies will serve as research coordinator.

#### 11. External Research Partnerships and funding

As indicated above, external research partnerships are considered essential to the activities of our research team. The investigators will apply to receive substantial financial support from the CIHR and from AllerGen (appendix D budget). The investigators will work closely with client organizations such as the Anaphylaxis Canada , AAIA ( allergy/Asthma Information Association ) , and the AQAA (Association québécoise des allergies alimentaires ). These support a cyber-society of people with food allergies and will provide support for our research activities from their limited budgets, again indicating the relevance of our research efforts to their needs.

| Name of Partner | Nature of participation | Contribution (CA\$) | Letter |
|-----------------|-------------------------|---------------------|--------|

| | | | | yes /no |
|--------------------|-----------|------|---------|---------|
| | | Cash | In-kind | |
| Anaphyalxis | | | 1000 | Y |
| Canada | | | | |
| AAIA | | | 1000 | Y |
| AQAA | | | 1000 | Y |
| Total value of par | tnerships | | | |

#### References

- (1) Decker WW, Campbell RL, Manivannan V, Luke A, St Sauver JL, Weaver A et al. The etiology and incidence of anaphylaxis in Rochester, Minnesota: a report from the Rochester Epidemiology Project. J Allergy Clin Immunol 2008; 122(6):1161-5.
- (2) Bohlke K, Davis RL, DeStefano F, Marcy SM, Braun MM, Thompson RS. Epidemiology of anaphylaxis among children and adolescents enrolled in a health maintenance organization. J Allergy Clin Immunol 2004; 113(3):536-42.
- (3) Sheikh A, Alves B. Hospital admissions for acute anaphylaxis: time trend study. BMJ 2000; 320(7247):1441.
- (4) Gold MS. EpiPen epidemic or good clinical practice? J Paediatr Child Health 2003; 39(5):376-7.
- (5) Liew WK, Williamson E, Tang ML. Anaphylaxis fatalities and admissions in Australia. J Allergy Clin Immunol 2009; 123(2):434-42.
- (6) Lin RY, Anderson AS, Shah SN, Nurruzzaman F. Increasing anaphylaxis hospitalizations in the first 2 decades of life: New York State, 1990 2006. Ann Allergy Asthma Immunol 2008; 101(4):387-93.
- (7) Gold MS, Sainsbury R. First aid anaphylaxis management in children who were prescribed an epinephrine autoinjector device (EpiPen). J Allergy Clin Immunol 2000; 106(1 Pt 1):171-6.
- (8) Simons FE, Roberts JR, Gu X, Simons KJ. Epinephrine absorption in children with a history of anaphylaxis. J Allergy Clin Immunol 1998; 101(1 Pt 1):33-7.

- (9) Plaut M, Sawyer RT, Fenton MJ. Summary of the 2008 National Institute of Allergy and Infectious Diseases-US Food and Drug Administration Workshop on Food Allergy Clinical Trial Design. J Allergy Clin Immunol 2009; 124(4):671-8.
- (10) Ben Shoshan M, Clarke AE. Anaphylaxis: past, present and future. Allergy 2010.
- (11) Garcia RR, Urra JM, Feo-Brito F, Galindo PA, Borja J, Gomez E et al. Oral rush desensitization to egg: efficacy and safety. Clin Exp Allergy 2011; 41(9):1289-96.
- (12) Buchanan AD, Green TD, Jones SM, Scurlock AM, Christie L, Althage KA et al. Egg oral immunotherapy in nonanaphylactic children with egg allergy. J Allergy Clin Immunol 2007; 119(1):199-205.
- (13) Itoh N, Itagaki Y, Kurihara K. Rush specific oral tolerance induction in school-age children with severe egg allergy: one year follow up. Allergol Int 2010; 59(1):43-51.
- (14) Zapatero L, Alonso E, Fuentes V, Martinez MI. Oral desensitization in children with cow's milk allergy. J Investig Allergol Clin Immunol 2008; 18(5):389-96.
- (15) Soller L, Ben-Shoshan M, Harrington DW, Knoll M, Fragapane J, Joseph L et al. Adjusting for nonresponse bias corrects overestimates of food allergy prevalence. J Allergy Clin Immunol Pract 2015; 3(2):291-3.
- (16) Byrne AM, Malka-Rais J, Burks AW, Fleischer DM. How do wee know when peanut and allergy have resolved, and how do we keep it resolved? Clin Exp Allergy 2010; 40(9):1303-11.
- (17) Hochstadter E, Clarke A, De SS, LaVieille S, Alizadehfar R, Joseph L et al. Increasing visits for anaphylaxis and the benefits of early epinephrine administration: A 4-year study at a pediatric emergency department in Montreal, Canada. J Allergy Clin Immunol 2016.
- (18) Bird JA, Feldman M, Arneson A, Dougherty I, Brown LS, Burk CM et al. Modified peanut oral immunotherapy protocol safely and effectively induces desensitization. J Allergy Clin Immunol Pract 2015; 3(3):433-5.
- (19) Pumphrey RS. Lessons for management of anaphylaxis from a study of fatal reactions. Clin Exp Allergy 2000; 30(8):1144-50.
- (20) McWilliam V, Koplin J, Lodge C, Tang M, Dharmage S, Allen K. The Prevalence of Allergy: A Systematic Review. Curr Allergy Asthma Rep 2015; 15(9):54.

- (21) Soller L, Ben-Shoshan M, Harrington DW, Knoll M, Fragapane J, Joseph L et al. Prevalence and predictors of food allergy in Canada: a focus on vulnerable populations. J Allergy Clin Immunol Pract 2015; 3(1):42-9.
- (22) Koppelman SJ, Wensing M, Ertmann M, Knulst AC, Knol EF. Relevance of Ara h1, Ara h2 and Ara h3 in peanut-allergic patients, as determined by immunoglobulin E Western blotting, basophil-histamine release and intracutaneous testing: Ara h2 is the most important peanut allergen. Clin Exp Allergy 2004; 34(4):583-90.
- (23) Roux KH, Teuber SS, Sathe SK.allergens. Int Arch Allergy Immunol 2003; 131(4):234-44.
- (24) Goetz DW, Whisman BA, Goetz AD. Cross-reactivity among edible nuts: double immunodiffusion, crossed immunoelectrophoresis, and human specific igE serologic surveys. Ann Allergy Asthma Immunol 2005; 95(1):45-52.
- (25) Ben Shoshan M, Harrington DW, Soller L, Fragapane J, Joseph L, St Pierre Y et al. A population-based study on peanut, tree nut, fish, shellfish, and sesame allergy prevalence in Canada. J Allergy Clin Immunol 2010; 125(6):1327-35.
- (26) Sampson HA, Ho DG. Relationship between food-specific IgE concentrations and the risk of positive food challenges in children and adolescents. J Allergy Clin Immunol 1997; 100(4):444-51.
- (27) Jones SM, Pons L, Roberts JL, Scurlock AM, Perry TT, Kulis M et al. Clinical efficacy and immune regulation with peanut oral immunotherapy. J Allergy Clin Immunol 2009; 124(2):292-300, 300.
- (28) Varshney P, Jones SM, Scurlock AM, Perry TT, Kemper A, Steele P et al. A randomized controlled study of peanut oral immunotherapy: clinical desensitization and modulation of the allergic response. J Allergy Clin Immunol 2011; 127(3):654-60.
- (29) Enrique E, Malek T, Pineda F, Palacios R, Bartra J, Tella R et al. Sublingual immunotherapy for hazelnut food allergy: a follow-up study. Ann Allergy Asthma Immunol 2008; 100(3):283-4.
- (30) Rolinck-Werninghaus C, Staden U, Mehl A, Hamelmann E, Beyer K, Niggemann B. Specific oral tolerance induction with food in children: transient or persistent effect on food allergy? Allergy 2005; 60(10):1320-2.
- (31) Jones SM, Burks AW, Keet C, Vickery BP, Scurlock AM, Wood RA et al. Long-term treatment with egg oral immunotherapy enhances sustained unresponsiveness that persists after cessation of therapy. J Allergy Clin Immunol 2016; 137(4):1117-27.

- (32) Blumchen K, Ulbricht H, Staden U, Dobberstein K, Beschorner J, de Oliveira LC et al. Oral peanut immunotherapy in children with peanut anaphylaxis. J Allergy Clin Immunol 2010; 126(1):83-91.
- (33) Vickery BP, Berglund JP, Burk CM, Fine JP, Kim EH, Kim JI et al. Early oral immunotherapy in peanut-allergic preschool children is safe and highly effective. J Allergy Clin Immunol 2017; 139(1):173-81.
- (34) Ballmer- Weber BK, Fernandez-Rivas M, Beyer K, Defernez M, Sperrin M, Mackie AR et al. How much is too much? Threshold dose distributions for 5 food allergens. J Allergy Clin Immunol 2015; 135(4):964-71.
- (35) Vadas P, Perelman B. Presence of undeclared peanut protein in chocolate bars imported from Europe. J Food Prot 2003; 66(10):1932-4.
- (36) Vickery BP. Low-Dose Oral Immunotherapy As an Early Intervention Strategy for Peanut Allergy. J Allergy Clin Immunol. 131[2], AB130. 1-2-0013.

Ref Type: Abstract

- (37) Sancho-Serra MC, Simarro M, Castells M. Rapid IgE desensitization is antigen specific and impairs early and late mast cell responses targeting FcepsilonRI internalization. Eur J Immunol 2011; 41(4):1004-13.
- (38) Turcanu V, Maleki SJ, Lack G. Characterization of lymphocyte responses to peanuts in normal children, peanut-allergic children, and allergic children who acquired tolerance to peanuts. J Clin Invest 2003; 111(7):1065-72.
- (39) Thottingal TB, Stefura BP, Simons FE, Bannon GA, Burks W, HayGlass KT. Human subjects without peanut allergy demonstrate T cell-dependent, TH2-biased, peanut-specific cytokine and chemokine responses independent of TH1 expression. J Allergy Clin Immunol 2006; 118(4):905-14.
- (40) Takayama N, Igarashi O, Keon MN, Kiyono H. Regulatory role of Peyer's patches for the inhibition of OVA-induced allergic diarrhea. Clin Immunol 2007; 123(2):199-208.
- (41) van Wijk F, Wehrens EJ, Nierkens S, Boon L, Kasran A, Pieters R et al. CD4+CD25+ T cells regulate the intensity of hypersensitivity responses to peanut, but are not decisive in the induction of oral sensitization. Clin Exp Allergy 2007; 37(4):572-81.
- (42) Cardoso CR, Teixeira G, Provinciatto PR, Godoi DF, Ferreira BR, Milanezi CM et al. Modulation of mucosal immunity in a murine model of foodinduced intestinal inflammation. Clin Exp Allergy 2008; 38(2):338-49.

- (43) Karlsson MR, Rugtveit J, Brandtzaeg P. Allergen-responsive CD4+CD25+ regulatory T cells in children who have outgrown cow's milk allergy. J Exp Med 2004; 199(12):1679-88.
- (44) Shreffler WG, Wanich N, Moloney M, Nowak-Wegrzen A, Sampson HA. Association of allergen-specific regulatory T cells with the onset of clinical tolerance to milk protein. J Allergy Clin Immunol 2009; 123(1):43-52.
- (45) Smith M, Tourigny MR, Noakes P, Thornton CA, Tulic MK, Prescott SL. Children with egg allergy have evidence of reduced neonatal CD4(+)CD25(+)CD127(lo/-) regulatory T cell function. J Allergy Clin Immunol 2008; 121(6):1460-6, 1466.
- (46) Schaub B, Liu J, Hoppler S, Haug S, Sattler C, Lluis A et al. Impairment of T-regulatory cells in cord blood of atopic mothers. J Allergy Clin Immunol 2008; 121(6):1491-9, 1499.
- (47) Torgerson TR, Linane A, Moes N, Anover S, Mateo V, Rieux-Laucat F et al. Severe food allergy as a variant of IPEX syndrome caused by a deletion in a noncoding region of the FOXP3 gene. Gastroenterology 2007; 132(5):1705-17.
- (48) Mori F, Bianchi L, Pucci N, Azzari C, De MM, Novembre E. CD4+CD25+Foxp3+ T regulatory cells are not involved in oral desensitization. Int J Immunopathol Pharmacol 2010; 23(1):359-61.
- (49) Tan TH, Ellis JA, Saffery R, Allen KJ. The role of genetics and environment in the rise of childhood food allergy. Clin Exp Allergy 2011.
- (50) Miller RL, Ho SM. Environmental epigenetics and asthma: current concepts and call for studies. Am J Respir Crit Care Med 2008; 177(6):567-73.
- (51) Lee DU, Agarwal S, Rao A. Th2 lineage commitment and efficient IL-4 production involves extended demethylation of the IL-4 gene. Immunity 2002; 16(5):649-60.
- (52) Jones B, Chen J. Inhibition of IFN-gamma transcription by site-specific methylation during T helper cell development. EMBO J 2006; 25(11):2443-52.
- (53) Tykocinski LO, Hajkova P, Chang HD, Stamm T, Sozeri O, Lohning M et al. A critical control element for interleukin-4 memory expression in T helper lymphocytes. J Biol Chem 2005; 280(31):28177-85.
- (54) Ben-Shoshan M, Kagan RS, Alizadehfar R, Joseph L, Turnbull E, St.Pierre Yvan et al. Is the prevalence of peanut allergy increasing? A five-year follow-up study on the prevalence of peanut allergy in primary school children in Montreal. Journal of Allergy and Clinical Immunology 123[4], 783-8. 2009.

Ref Type: Journal (Full)

- (55) Hourihane JO, Kilburn SA, Dean P, Warner JO. Clinical characteristics of peanut allergy. Clin Exp Allergy 1997; 27(6):634-9.
- (56) Brown SG. Clinical features and severity grading of anaphylaxis. J Allergy Clin Immunol 2004; 114(2):371-6.
- (57) Sicherer SH, Burks AW, Sampson HA. Clinical features of acute allergic reactions to peanut and tree nuts in children. Pediatr 1998; 102(1):e6.
- (58) Bindslev-Jensen C, Ballmer-Weber BK, Bengtsson U, Blanco C, Ebner C, Hourihane J et al. Standardization of food challenges in patients with immediate reactions to foods--position paper from the European Academy of Allergology and Clinical Immunology. Allergy 2004; 59(7):690-7.
- (59) Perry TT, Matsui EC, Conover-Walker MK, Wood RA. Risk of oral food challenges. J Allergy Clin Immunol 2004; 114(5):1164-8.
- (60) Calvani M, Sopo SM. Exercise-induced anaphylaxis caused by wheat during specific oral tolerance induction. Ann Allergy Asthma Immunol 2007; 98(1):98-9.
- (61) Caminiti L, Passalacqua G, Vita D, Ruggeri P, Barberio G, Pajno GB. Food-exercise-induced anaphylaxis in a boy successfully desensitized to cow milk. Allergy 2007; 62(3):335-6.
- (62) Wedi B, Novacovic V, Koerner M, Kapp A. Chronic urticaria serum induces histamine release, leukotriene production, and basophil CD63 surface expression--inhibitory effects of anti-inflammatory drugs. J Allergy Clin Immunol 2000; 105(3):552-60.
- (63) Gentinetta T, Pecaric-Petkovic T, Wan D, Falcone FH, Dahinden CA, Pichler WJ et al. Individual IL-3 priming is crucial for consistent in vitro activation of donor basophils in patients with chronic urticaria. J Allergy Clin Immunol 2011.
- (64) Gyimesi E, Sipka S, Danko K, Kiss E, Hidvegi B, Gal M et al. Basophil CD63 expression assay on highly sensitized atopic donor leucocytes-a useful method in chronic autoimmune urticaria. Br J Dermatol 2004; 151(2):388-96.
- (65) Flokstra-de Blok BM, Dubois AE. Quality of life in food allergy: valid scales for children and adults. Curr Opin Allergy Clin Immunol 2009; 9(3):214-21.

- (66) Saleh-Langenberg J, Goossens NJ, Flokstra-de Blok BM, Kollen BJ, van der Meulen GN, Le TM et al. Predictors of health-related quality of life of European food-allergic patients. Allergy 2015; 70(6):616-24.
- (67) Shertzer CL, Lookingbill DP. Effects of relaxation therapy and hypnotizability in chronic urticaria. Arch Dermatol 1987; 123(7):913-6.
- (68) Skripak JM, Nash SD, Rowley H, Brereton NH, Oh S, Hamilton RG et al. A randomized, double-blind, placebo-controlled study of milk oral immunotherapy for cow's milk allergy. J Allergy Clin Immunol 2008; 122(6):1154-60.
- (69) Caminiti L, Passalacqua G, Barberi S, Vita D, Barberio G, De Luca R et al. A new protocol for specific oral tolerance induction in children with IgE-mediated cow's milk allergy. Allergy Asthma Proc 2009; 30(4):443-8.
- (70) Martorell A, De la Hoz B, Ibanez MD, Bone J, Terrados MS, Michavila A et al. Oral desensitization as a useful treatment in 2-year-old children with cow's milk allergy. Clin Exp Allergy 2011; 41(9):1297-304.
- (71) Fernandez-Rivas M, Garrido FS, Nadal JA, Diaz dD, Garcia BE, Gonzalez-Mancebo E et al. Randomized double-blind, placebo-controlled trial of sublingual immunotherapy with a Pru p 3 quantified peach extract. Allergy 2009; 64(6):876-83.
- (72) Vassallo MF, Banerji A, Rudders SA, Clark S, Mullins RJ, Camargo CA, Jr. Season of birth and food allergy in children. Ann Allergy Asthma Immunol 2010; 104(4):307-13.
- (73) Pali-Scholl I, Jensen-Jarolim E. Anti-acid medication as a risk factor for food allergy. Allergy 2010.
- (74) Gourbeyre P, Denery S, Bodinier M. Probiotics, prebiotics, and synbiotics: impact on the gut immune system and allergic reactions. J Leukoc Biol 2011; 89(5):685-95.
- (75) Poole JA, Barriga K, Leung DY, Hoffman M, Eisenbarth GS, Rers M et al. Timing of initial exposure to cereal grains and the risk of wheat allergy. Pediatrics 2006; 117(6):2175-82.
- (76) Du Toit G, Katz Y, Sasieni P, Mesher D, Maleki SJ, Fisher HR et al. Early consumption of peanuts in infancy is associated with a low prevalence of peanut allergy. J Allergy Clin Immunol 2008; 122(5):984-91.
- (77) Katz Y, Rajuan N, Goldberg MR, Eisenberg E, Heyman E, Cohen A et al. Early exposure to cow's milk protein is protective against IgE-mediated cow's milk protein allergy. J Allergy Clin Immunol 2010; 126(1):77-82.

- (78) Joseph CL, Ownby DR, Havstad SL, Woodcroft KJ, Wegienka G, Mackechnie H et al. Early complementary feeding and risk of food sensitization in a birth cohort. J Allergy Clin Immunol 2011.
- (79) Koplin JJ, Osborne NJ, Wake M, Martin PE, Gurrin LC, Robinson MN et al. Can early introduction of egg prevent egg allergy in infants? A population-based study. J Allergy Clin Immunol 2010; 126(4):807-13.
- (80) DesRoches A, Infante-Rivard C, Paradis L, Paradis J, Haddad E. Peanut allergy: is maternal transmission of antigens during pregnancy and breastfeeding a risk factor? J Investig Allergol Clin Immunol 2010; 20(4):289-94.
- (81) Sicherer SH, Wood RA, Stablein D, Lindblad R, Burks AW, Liu AH et al. Maternal consumption of peanut during pregnancy is associated with peanut sensitization in atopic infants. J Allergy Clin Immunol 2010; 126(6):1191-7.
- (82) Chung SY, Butts CL, Maleki SJ, Champagne ET. Linking peanut allergenicity to the processes of maturation, curing, and roasting. J Agric Food Chem 2003; 51(15):4273-7.
- (83) Liu GM, Cheng H, Nesbit JB, Su WJ, Cao MJ, Maleki SJ. Effects of boiling on the IgE-binding properties of tropomyosin of shrimp (Litopenaeus vannamei). J Food Sci 2010; 75(1):T1-T5.
- (84) Samson KT, Chen FH, Miura K, Odajima Y, Iikura Y, Naval RM et al. IgE binding to raw and boiled shrimp proteins in atopic and nonatopic patients with adverse reactions to shrimp. Int Arch Allergy Immunol 2004; 133(3):225-32.
- (85) Milner JD, Stein DM, McCarter R, Moon RY. Early infant multivitamin supplementation is associated with increased risk for food allergy and asthma. Pediatrics 2004; 114(1):27-32.
- (86) Camargo CA, Jr., Clark S, Kaplan MS, Lieberman P, Wood RA. Regional differences in EpiPen prescriptions in the United States: the potential role of vitamin D. J Allergy Clin Immunol 2007; 120(1):131-6.
- (87) Mullins RJ, Clark S, Camargo Jr CA. Regional variation in infant hypoallergenic formula prescriptions in Australia. Pediatr Allergy Immunol 2009.
- (88) Mullins RJ, Clark S, Camargo CA, Jr. Regional variation in epinephrine autoinjector prescriptions in Australia: more evidence for the vitamin D-anaphylaxis hypothesis. Ann Allergy Asthma Immunol 2009; 103(6):488-95.

# Appendix A: Disease burden and gaps.

Table 2. Primary and secondary prevention measures for food allergies<sup>a</sup>

| Primary | Route of | Reference number | Secondary pr |
|---|---|---|---|
| prevention | desensitization | | |
| | PO, SL | (14;68-70) | Avoidance of |
| Tree nut | PO | (11-13) | education of alle |
| Peanut | PO | (27) | their care-givers |
| Tree nut | SL | (29) | avoidance, impro |
| Peach | SL | (71) | prepackaged foo |
| | | | wearing of Medi |
| | | | specific food alle |
| | Tree nut Peanut Tree nut | prevention desensitization PO, SL Tree nut PO Peanut PO Tree nut SL | prevention desensitization PO, SL (14;68-70) Tree nut PO Peanut PO Tree nut SL (29) |

<sup>&</sup>lt;sup>a</sup> only the most common foods, drugs and insect desensitization approaches are

mentioned.

PO, Per os; SL, Sublingual; SC,

Table 2.Environmental factors associated with food allergy.

| Factor | study | Type of study | Effect |
|--------|-------|---------------|--------|

| Season | Vassall | Case control | Children younger than 5 years born in fall or winter had |
|---|---|---|---|
| | o MF | | higher odds of food allergy compared with controls. |
| Drugs | Palli- | Case control | The relative risk to develop food-specific IgE after anti- |
| | Scholl | | therapy was 10.5 (95% CI,1.44,76.48). |
| Microbial | Gourbe | Review of case | No clear conclusion regarding probiotic beneficial effec |
| exposure | yre | control and cohort | the prevention or treatment of allergy . |
| | | studies | |
| Food | Poole | Cohort | After adjusting for breastfeeding duration, introduction |
| consumption | JA | | cereal, family history of allergy, and history of food allergy |
| (quantity | | | 6 months of age, age at initial exposure to cereal grains cor |
| and timing) | | | to be strongly associated with wheat allergy (≥7 months: ac |
| | | | OR: 3.8; 95% CI, 1.18,12.28) |
| | Du Toit | Case control | After adjustment for atopy, other food allergies, age, and |
| | | | the RR for peanut allergy in the UK vs Israel is 5.8 (95% C |
| | | | 2.8,11.8), and largest and most significant difference in an |
| | | | between the UK and Israel was observed in the age of intro |
| | | | of peanut (P < .0001). By 9 months of age, 69% of Israelis |
| | | | eating peanut compared with only 10% of UK infants. |
| | Katz | Cohort | The OR was 19.3 (95% CI, 6.0,62.1) for development o |
| | | | mediated CMA among infants with exposure to cow prote |
| | | | age of 15 days or more ( $P < .001$ ) vs those introduced to co |
| | | | protein before 15 days. |

| | Joseph | Cohort | Early feeding reduced the risk of peanut sensitization an |
|---|---|---|---|
| | | | children with a parental history [adjusted OR, 0.2 (95% CI |
| | | | 0.1,0.7); P = .007]. The relationship also became significan |
| | | | forwhen a cutoff for IgE of ≥0.70 IU/mL was used [adjusted] |
| | | | 0.5 (95% CI, 0.3,0.9)]. |
| | Koplin | Case control | Introduction of cooked at age 4 to 6 months, vs later exp |
| | | | reduced the risk of allergy [OR, 0.2 (95% CI, 0.06-0.71)]. |
| | Des | Case control | The reported consumption of peanuts during pregnancy |
| | Roches | | breastfeeding was higher in the case group (those who deve |
| | | | peanut allergy and associated with an increased risk of pea |
| | | | allergy in offspring [OR, 4.22 (95%CI, 1.57,11.30) and OR |
| | | | (95% CI, 1.31,3.97) for pregnancy and breastfeeding, |
| | | | respectively]. |
| | Sichere | Case control | Multivariate analysis including clinical, laboratory, and |
| | r | | demographic variables showed frequent peanut consumption |
| | | | during pregnancy {OR, 2.9(95% CI, 1.7,4.9)] to be associated |
| | | | with peanut IgE ≥5 kUA/L. |
| Food | Chung | Laboratory | After curing and roasting, mature peanuts exhibited |
| processing | | analysis | approximately 20% higher levels of advanced glycation en |
| | | | adducts and higher IgE binding vs immature peanuts. |
| | Yadzir | Laboratory | Extracts from raw shrimp bound higher IgE than extract |
| | | analysis | boiled shrimp, but the purified boiled tropomysoin (the ma |
| | | | shrimp allergen) demonstrates higher IgE binding vs raw si |

| | Samson | Laboratory | Thermal processing can lead to the formation of new an |
|---|---|---|---|
| | | analysis | structures. |
| Vitamin | Milner | Cohort | Early vitamin D use (within the first 6 months of life) w |
| D | | | associated with a higher risk for food allergies in the exclusion |
| | | | formula-fed population [OR,1.63( 95% CI,1.21,2.20)]. Vita |
| | | | use at 3 years of age was associated with increased risk for |
| | | | allergies but not asthma in both breastfed [OR,1.62(95% |
| | | | CI,1.19,2.21) ]and exclusively formula-fed infants [OR, 1.1 |
| | | | CI,1.03,1.88)]. |
| | Cramag | Ecologic study | Strong north-south gradient for the prescription of EpiPo |
| | o | | the United States, with the highest rates found in New Eng |
| | | | [adjusted $\beta$ for New England vs the rest of the US, 4.07 (95) |
| | | | 2.77,5.36)] |
| | Mulins | Ecologic study | Using multivariate analysis, EpiPen prescription rates t |
| | et al | | higher in southern latitudes (less sunlight) compared with r |
| | | | regions [β, -19.22( 95% CI, -26.71 , -11.73)]. |
| | Mulins | Ecologic study | Southern latitudes were associated with higher hypoalle |
| | et al | | formulae prescription rates [beta, -147.98( 95% CI,-281.83 |
| | | | 14.14)]. |

OR, odds ratio;RR, Relative Risk; CI,confidence interval ;CMA, Cow's Allergy

Appendix B. protocols.

A1. BPCFC

Double-blind, placebo-controlled food challenge (BPCFC) up to 100 mg (144 mg cumulative)done at screening and 3 months post OIT

| Dose | Cumulative |
|--------|------------|
| 1 mg | 1 mg |
| 3 mg | 4 mg |
| 10 mg | 14 mg |
| 30 mg | 44 mg |
| 100 mg | 144 mg |
| 300 | 444 |

A 2. Scale for Grading Reaction Severity

| Score Symptom | Action |
|---------------|--------|
|---------------|--------|

| Mild | Pruritus, | Observe |
|---|---|---|
| | Urticaria, | May give Antihistamine (e.g. |
| | Flushing, | Benadryl or Reactin as prescribed |
| | Rhinoconjunctivitis | Call Research Team |
| | | Research team will evaluate if dose |
| | | adjustment is needed and if next dose |
| | | will be given at home or in hospital. |
| Moderate | Angioedema, | Give epinephrine IM as per protocol |
| | Throat tightness, | Give Antihistamine (e.g. Benadryl or |
| | Gastrointestinal complaints (cramping, | Reactin as prescribed |
| | . pain,vomiting,diarrhea) | Seek urgent care (hospital emergency |
| | Respiratory symptoms (Cough, Mucous | room) |
| | production) | Call Research team |
| | | To give next adjusted dose in hospital |
| | | research unit (CIM) |
| Severe | Wheeze, Respiratory Distress | Give epinephrine IM as per protocol |
| | Hypoxia, | Give Antihistamine (e.g. Benadryl or |
| | Cyanosis, | Reactin as prescribed |
| | Hypotension | Call 911 |
| | Circulatory collapse (Shock) | Seek urgent care (transfer to hospital |
| | | emergency room) |
| | | Call Research team; if the symptoms |
| | | are not improving within 10 minutes |
| | | of the first dose, instructions will be |
| | | given from the team regarding use of |
| | | a second dose of epinephrine. |

# B1. Initial Escalation: Day 1 and 2

- Verify no wheezing, flare of atopic disease, or other intercurrent illness
- Update history and con meds
- Vital signs and PE
- PEFR
- Dose escalation at 20 minute intervals
- Post-dose vital signs

- Vital signs q30min x3 post last dose
- Monitoring for AEs (see

| Day 1 | Day 1 | Day 2 | Day 2 |
|---|---|---|---|
| Dose ( raw | Dose ( crushed | Dose( raw peanut/ | Dose( crushed raw |
| peanut/ tree nut) | peanut/ tree nut) | tree nut protein) | peanut/ tree nut) |
| 0.5mg | 2.0 mg | 3mg | |
| 1mg | 4.0 mg | | |
| 1.5mg | 6.0 mg | | |
| 2.5 mg | 10.0 mg | | |
| 3mg | 12 mg | | |
| 3.5mg | 14 mg | | |
| 4mg | 16 mg | | |
| 4.5mg | 18 mg | | |
| 5mg | 20 mg | | |

# B2a. Build up phase for 300mg (group A)

| | <u> </u> | D. | | |
|---|---|---|---|---|
| | Dose | Dose | | |
| | (peanut/tree | (crushed | | Percent |
| | nut protein) | peanut/tree nut | Interval | Increase from |
| Dose Number | (mg) | (mg) | (weeks) | <b>Previous Dose</b> |

| 1 | 3 | | 2 | |
|----|-----|--------------------|-------|------|
| 2 | 6 | 24 | 2 | 100% |
| 3 | 12 | 48 | 2 | 100% |
| 4 | 20 | 80 | 2 | 67% |
| 5 | 40 | 160 | 2 | 100% |
| 6 | 80 | 320 | 2 | 100% |
| 7 | 120 | 480 | 2 | 50% |
| 8 | 160 | 640 | 2 | 33% |
| 9 | 200 | 800 | 2 | 25% |
| 10 | 240 | 960 | 2 | 20% |
| 11 | 300 | 1200 | Enter | 25% |
| ** | 200 | Maintenance Period | | |

B2a. Build up phase for 30mg (group B)

| | Dose | Dose | | |
|-------------|-------------|-----------------|----------|---------------|
| | peanut/tree | crushed | | Percent |
| | nut protein | peanut/tree nut | Interval | Increase from |
| Dose Number | (mg) | (mg) | (weeks) | Previous Dose |
| 1 | 3 | 12 | 2 | |

| 2 | 6 | 24 | 2 | 100% |
|----|----|-----|----------------|-------|
| 3 | 12 | 48 | 2 | 100% |
| 4 | 20 | 80 | 2 | 67% |
| 5 | 30 | 120 | 2 | 50% |
| 6 | 30 | 120 | 2 | 00% |
| 7 | 30 | 120 | 2 | 0% |
| 8 | 30 | 120 | 2 | 0% |
| 9 | 30 | 120 | 2 | 0% |
| 10 | 30 | 120 | 2 | 0% |
| 11 | 30 | 120 | Enter | 0% |
| 11 | 30 | | Maintenance Pe | eriod |

If the subject does not tolerate a given dose and symptoms are mild, then that dose or the previously tolerated one is repeated, and the protocol proceeds as outlined. If the subject experiences significant symptoms, then the protocol is stopped, and the highest tolerated dose is used as the starting daily dose.

All doses will be pre-weighed and encapsulated to blind both patients and evaluating physicians

After achieving a dose of 300 mg(group A) or 30 mg (group B), the subject will return for a first maintenance visit 2 weeks later.

• Visits are then every 4 weeks until Exit Visit

# B3. Challenges during maintenance period ( for group A or B):

| Dose | Dose | Cumulative | Cumulative |
|------------------|------------------|------------------|------------------|
| (peanut protein) | (crushed peanut) | (peanut protein) | (crushed peanut) |
| 3 mg | 12 mg | 3 mg | 12 mg |
| 10 mg | 40 mg | 13 mg | 52 mg |
| 30 mg | 120 mg | 43 mg | 172 mg |
| 100 mg | 400 mg | 143 mg | 572 mg |
| 300 mg | 1200 mg | 443 mg | 1772 mg |
| 600 mg | 2400 mg | 1043 mg | 4172 mg |
| 1000 mg | 4000 mg | 2043 mg | 8172 mg |

Appendix C. Budget

Total budget estimate: 78,000CAD per year including:

| | Estimate (CAD) | comment |
|--------------------------------------|----------------|--------------------|
| Yearly salary for an | 35,000 | |
| undergraduate student for salary | | |
| that will support training in Lab | | |
| evaluation mechanisms for | | |
| tolerance detection | | |
| Study coordinator | 40,000 | Yearly salary with |
| | | benefits |
| Paediatric test center (70CAD | 3000 | |
| for each blood sample) | | |
| Staining with monoclonal Abs | 3000 | |
| Use of FACS | 3000 | |
| CBA | 3500 | |
| Culture materials and stimulating | 3500 | |
| material | | |
| Travel expenses for presentation | 5000 | |
| of results in scientific conferences | | |
| | 78,000 | yearly |

Appendix D: Flow chart of study procedures

